CLINICAL TRIAL: NCT05377086
Title: Comparison of the Effectiveness of the Structured 3D Exercise and the Conventional Exercise Program for Scoliosis in Children With Rheumatic Disease
Brief Title: Structured 3D Exercise and the Conventional Exercise Program for Scoliosis in Children With Rheumatic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Eylül Pınar KISA, Lecturer, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHD Thesis
Record Dates: First submitted 2022-05-01; First posted 2022-05-17 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Scoliosis; Juvenile Idiopathic Arthritis
Keywords: scoliosis; Juvenile idiopathic arthritis; 3D exercise
MeSH Terms: conditions — Scoliosis; Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- schroth group (Experimental): This arm was planned as the exercise group which includes Schroth 3-Dimensional scoliosis exercise.
  Interventions: Other: Schroth 3-Dimensional scoliosis exercise
- conventional group (Experimental): This arm was planned as the exercise group which includes conventional scoliosis exercise.
  Interventions: Other: conventional scoliosis exercise

INTERVENTIONS:
Other: Schroth 3-Dimensional scoliosis exercise — Schroth 3-Dimensional scoliosis exercises
  Arms: schroth group
Other: conventional scoliosis exercise — conventional scoliosis exercise
  Arms: conventional group

SUMMARY:
Usage including cases followed up with rheumatism diagnosis and treatment in Istanbul University-Cerrahpasa Medical Faculty Pediatric Rheumatology Clinic, Physiotherapy and Rehabilitation Unit. The study included 50 patients with a spinal x-ray scoliosis problem, aged 8-16 years, who were diagnosed with rheumatism at least 6 months ago, whose medical treatment was stable, Risser 0-4 and exercise indication (Cobb = 10-45ͦ). Patients with additional neurological diagnosis against rheumatism, who have received any previous treatment for a spine problem, who have a mental state and who do not have the consent of their family will not be included. The cases will be divided into 2 groups by method. In the first group (n = 25), structured 3-dimensional scoliosis exercises are taught in the clinic, and the second group (n = 25) is taught conventional physiotherapy applications (posture-core applications-bennet protocols) in the clinic, and both groups are followed by the WTE method.

DETAILED DESCRIPTION:
The demographic and clinical characteristics of all subjects willing to participate in the study will be questioned with the "Sociodemographic Data Form". Sociodemographic data form; pain, age, gender, height, weight, type of rheumatism, how many years ago the patient was diagnosed, the presence of rheumatism and scoliosis in the family, the drugs used, exercise habits, exacerbation history, whether they used a device before, and the awareness of the family about scoliosis. The trunk rotation angles with the forward bend test and the Cobb angle with the SubrotoAngleAid application via x-ray. Respiratory functions will be evaluated with portable spirometer, body awareness will be evaluated with Walter Reed Visual Assessment Scale, and quality of life will be evaluated with Scoliosis Research Association Scale-22 (SRS-22). After the evaluations, in the first treatment session in the clinic, the cases in the first group; Body awareness, respiratory control, differences between rotational and normal breathing, posture exercises and core stabilization exercises will be taught and family training will be provided. In the next session, a home program will be created by applying 3D scoliosis exercises that are structured according to the needs of the patients. Body awareness, respiratory control, posture exercises and core stabilization exercises will be taught and family training will be given to the patients in the second group in the first treatment session. In the next session, conventional exercises for the needs of the cases will be taught and a home exercise program will be created. Both groups will be interviewed for 2-week periods using the WTE method, and the exercises will be progressed gradually as needed. At the beginning of the treatment and in the 6th month, all evaluations will be repeated and the effectiveness of the exercises will be investigated. SPSS (Statistical Package for Social Sciences) (SPSS 21.0) statistical program will be used in the statistical analysis of the data. In all statistical analyzes, p <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Cases with a diagnosis of rheumatism in whom scoliosis problems were detected by spine X-ray,
* be between the ages of 8-16,
* Being between 0-4 in the riser,
* Being in exercise indication (Cobb=10-45 ˚)

Exclusion Criteria:

* Having an additional neurological or orthopedic diagnosis other than scoliosis accompanying rheumatism and affecting treatment results
* Having had any surgery on the spine
* Have had previous scoliosis treatment poor mental state

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Cobb angle | 0-6 month
  Measuring the scoliosis angle on x-ray is the most commonly used method. The Cobb angle is most commonly used to measure the magnitude of the curve. Measurements are made on a standing posteroanterior spine radiograph as standard. To determine the boundaries of the scoliosis, a line is drawn parallel to the upper line of the vertebra with the greatest deviation. Similarly, for the lower border, a line is drawn parallel to the lowest vertebra. Vertical lines are drawn parallel to these two lines and the angle between the two lines is measured. This angle is defined as the scoliosis angle (Cobb angle). Radiological imaging will only be applied to children who are considered to be in need by the doctor as a result of physical examination. The measurement of the Cobb angle will be made on the X-ray via the SubrotoAngleAid application.
Trunk rotation with Scoliometer | 0-6 month
  The trunk rotation angle will be measured with a scoliometer. It is an easy to use, reliable, practical and specially designed inclinometer in the clinical evaluation of scoliosis. It is accepted as a clinical evaluation method used in addition to radiological methods in determining the efficacy of treatment and the prognosis of scoliosis.

SECONDARY OUTCOMES:
Physical deformity assesment using with The Walter Reed Visual Assessment Scale (WRVAS) | 0-6 month
  The Walter Reed Visual Assessment Scale (WRVAS) developed to evaluate the physical deformity perceived by patients with idiopathic scoliosis. Walter Reed Visual Evaluation Scale evaluates deformity from 7 aspects; spine curvature, rib protrusion, lumbar protrusion, thorax deformity relative to pelvis (alignment disorder), trunk imbalance, shoulder and scapula asymmetry. For each of the 7 questions that make up the Walter Reed visual assessment scale, there is an answer section consisting of 5 different pictures indicating different degrees of deformity. Each deformity is scored with these pictures as a minimum of "1" and a maximum of "5". The scale will be filled in by the therapist.
FEV1 | 0-6 month
  It is a physiological test in which the volume of air an individual inhales or exhales is evaluated as a function of time. Pulmonary function test will be done with a portable spirometer (Contec SP10W). Forced expiration test; calm breathing followed by a forced inspiration followed by an expiration as fast and deep (forced) as possible. During the test, the patient will be placed in a sitting position in a way that is comfortable and the patient will be prevented from breathing in and out of the nose with the nose clip. Maneuvers that may affect the test results such as bending forward and neck flexion during forced expiration will be prevented. Expiration should continue for at least six seconds and eventually plateau. Care will be taken to ensure that there is no leakage in the system.
FVC | 0-6 month
  It is a physiological test in which the volume of air an individual inhales or exhales is evaluated as a function of time. Pulmonary function test will be done with a portable spirometer (Contec SP10W). Forced expiration test; calm breathing followed by a forced inspiration followed by an expiration as fast and deep (forced) as possible. During the test, the patient will be placed in a sitting position in a way that is comfortable and the patient will be prevented from breathing in and out of the nose with the nose clip. Maneuvers that may affect the test results such as bending forward and neck flexion during forced expiration will be prevented. Expiration should continue for at least six seconds and eventually plateau. Care will be taken to ensure that there is no leakage in the system.
PEF | 0-6 month
  It is a physiological test in which the volume of air an individual inhales or exhales is evaluated as a function of time. Pulmonary function test will be done with a portable spirometer (Contec SP10W). Forced expiration test; calm breathing followed by a forced inspiration followed by an expiration as fast and deep (forced) as possible. During the test, the patient will be placed in a sitting position in a way that is comfortable and the patient will be prevented from breathing in and out of the nose with the nose clip. Maneuvers that may affect the test results such as bending forward and neck flexion during forced expiration will be prevented. Expiration should continue for at least six seconds and eventually plateau. Care will be taken to ensure that there is no leakage in the system.
QUALITY OF LIFE ASSESSMENT | 0-6 month
  Scoliosis Research Society Scale-22 (SRS-22)" questionnaire is an inquiry form designed for scoliosis and evaluating quality of life. It consists of 23 questions with five subgroups. These subgroups are; pain, image/appearance, function/activity, mental health, and treatment satisfaction. It is defined as 0 (worst) and 5 (best) points for each question. Patients will be asked to mark the answers that are suitable for them and the form will be filled. (because of pandemic, its not completed)

CONTACTS AND LOCATIONS:
Locations (1):
- Eylül Pınar Kısa, Istanbul, Turkey (Türkiye)